CLINICAL TRIAL: NCT01773486
Title: An Exploratory Study to Evaluate the Ability of the Citrus Polyphenol Hesperidin to Improve Insulin Sensitivity in Healthy Subjects and to Ameliorate Insulin Resistance in Obese Subjects
Brief Title: Effects of Hesperidin on Insulin Sensitivity
Acronym: EHIS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not funded
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Kashif Munir, Assistant Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00051658
Record Dates: First submitted 2013-01-17; First posted 2013-01-23 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Obesity; Insulin Resistance
Keywords: Obesity; Insulin Resistance; Endothelial dysfunction; Blood pressure
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Hesperidin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hesperidin (Active Comparator): Subjects will receive oral hesperidin 500 mg/day
  Interventions: Drug: Hesperidin
- Placebo (Placebo Comparator): subjects will receive matching placebo to hesperidin daily for 1 month
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hesperidin — Citrus polyphenol, hesperidin
  Arms: Hesperidin
Drug: Placebo — Placebo matching hesperidin
  Arms: Placebo

SUMMARY:
This study will examine whether hesperidin, a major component of citrus fruits, affects how the body responds to insulin in healthy and obese people. Laboratory studies suggest that hesperidin treatment lowers blood pressure, lowers blood sugar and increases blood flow. This study will see if hesperidin improves insulin resistance or insulin's effects on blood flow in people with insulin resistance.

Healthy normal weight or overweight people between 21 and 65 years of age may be eligible for this study. Participants are randomly assigned to take hesperidin or a placebo (inactive dummy pill ) for a 4-week treatment phase.

DETAILED DESCRIPTION:
This study will examine whether hesperidin, a major component of citrus fruits, affects how the body responds to insulin in healthy and obese people. Insulin is not as effective in people who are overweight, have high blood pressure or diabetes. This condition is known as insulin resistance. Laboratory studies suggest that hesperidin treatment lowers blood pressure, lowers blood sugar and increases blood flow. This study will see if hesperidin improves insulin resistance or insulin's effects on blood flow in people with insulin resistance.

Healthy normal weight or overweight people between 21 and 65 years of age may be eligible for this study. Participants are randomly assigned to take hesperidin or a placebo (inactive dummy pill ) for a 4-week treatment phase. In addition to treatment, participants undergo the following procedures during the study period:

Screening, including medical history, physical examination and blood and urine tests.

Complete a dietary and physical activity questionnaire and consult with a dietitian

Blood and urine tests

At-home and clinic blood pressure monitoring

Glucose clamp test to measure how the body responds to insulin. This test is done two times during the study. A needle is placed in a vein in each of the subject's arms, one for sampling blood and the other for infusing insulin, glucose and potassium. Glucose and insulin levels, electrolytes, lipids, fatty acids, cytokines and hesperidin levels are measured. We will also use tracer-labeled glucose to determine how much glucose the body produces in the fasting state and during the clamp. This type of glucose has low levels of radiation.

Forearm blood flow measurement with finger plethysmography device. Before beginning the glucose clamp test, a test of how well the blood vessels relax is done. A device that measures the blood flow in the vessels of the forefingers is used. The test is performed at the before the glucose clamp test and again 2 hours after the beginning of the clamp.

ELIGIBILITY:
Inclusion Criteria:

Healthy Subjects - Men and women in good general health with no significant underlying illnesses who are between the ages of 21 - 65 years of age with HbA1C < 5.7 %, fasting blood glucose < 100 mg/dL, blood pressure less than 120/80, and BMI between 20 - 25 kg/m2. Subjects should have never smoked tobacco or not smoked within the previous year.

Obese Subjects - Men and women in good general health with no significant underlying illnesses except obesity who are between the ages of 21 - 65 years of age with HbA1C < 5.7 %, fasting blood glucose < 100 mg/dl, blood pressure less than 130/90, and BMI between 30 - 45 kg/m2.

Exclusion Criteria:

* Subjects will be excluded from our study if they are pregnant, breastfeeding, or if they plan pregnancy prior to the end of the study. In addition, subjects will be excluded if their age > 65 yrs, BMI ≥ 45 kg/m2, or have liver disease (including liver transaminase levels greater than twice the upper limit of normal), pulmonary disease, renal insufficiency (serum creatinine greater than 2.0 mg/dl), coronary heart disease, heart failure (New York Heart Association heart failure Class III or IV), peripheral vascular disease, coagulopathy, Major depressive disorder, actively smoking or used tobacco within last year, history of cancer, in treatment for any form of cancer, positive tests for HIV, hepatitis B or C, or take systemic corticosteroids, thiazolidinediones (within 3 months), insulin, or anticoagulants, use food supplements that cannot be discontinued, regular intake of 8 or more cups of tea per week within 3 months prior to study entry, regular alcoholic beverage intake of more than two drinks per day (a drink corresponds to approximately 12 ounces of beer, 4 ounces of table wine, and between 1 and 1.5 ounces of 80-proof spirits), poor compliance during run-in period or regular use of medications that affect insulin sensitivity, blood pressure or vascular function and that cannot be discontinued. In addition, history of any other medical disease, laboratory abnormalities, or psychological conditions that would make the subject (based upon the principal investigator's judgment) unsuitable for study enrollment. Subjects will be excluded if they are unable to give informed consent for all procedures.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity (determined by glucose clamp) | 1 month
  To determine if oral hesperidin consumption (500 mg p.o. daily for 1 month) improves insulin sensitivity (determined by glucose clamp) in healthy individuals or improves insulin resistance in subjects with obesity when compared with placebo treatment

SECONDARY OUTCOMES:
basal hepatic glucose production | 1 month
  Determine whether or not hesperidin treatment reduces basal hepatic glucose production in obese and lean subjects using tracer-labeled glucose.
endothelial function | 1 month
  Determine if oral hesperidin consumption (500 mg p.o. daily for 1 month) improves baseline and insulin-stimulated endothelial function as measured by finger plethysmography via Endo-PAT (before and during glucose clamp studies)
blood pressure | 1 month
  Determine if oral hesperidin treatment reduces systolic and/or diastolic blood pressure in obese and lean subjects.
Inflammatory markers | 1 month
  Determine if oral hesperidin consumption (500 mg p.o. daily for 1 month) alters plasma levels of pro- and anti-inflammatory cytokines

OTHER OUTCOMES:
pharmacokinetics | 1 month
  Determine steady-state levels of hesperidin before and after 1 month treatment with hesperidin or placebo. Determine hesperidin pharmacokinetics in plasma after oral administration of hesperidin (500 mg)

CONTACTS AND LOCATIONS:
Overall Officials: Kashif Munir, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

REFERENCES:
- [Background] Rizza S, Muniyappa R, Iantorno M, Kim JA, Chen H, Pullikotil P, Senese N, Tesauro M, Lauro D, Cardillo C, Quon MJ. Citrus polyphenol hesperidin stimulates production of nitric oxide in endothelial cells while improving endothelial function and reducing inflammatory markers in patients with metabolic syndrome. J Clin Endocrinol Metab. 2011 May;96(5):E782-92. doi: 10.1210/jc.2010-2879. Epub 2011 Feb 23. PMID 21346065